CLINICAL TRIAL: NCT01207505
Title: Emotion Regulation Group Therapy for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thilo Deckersbach, Director of Psychology, Bipolar Clinic and Research Program Associate Professor of Psychology, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-001083
Record Dates: First submitted 2010-09-07; First posted 2010-09-23 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Bipolar I Disorder
Keywords: bipolar disorder; depression; mania; emotion regulation; dialectical behavior therapy; group therapy; mindfulness
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enchancing Emotion Regulation (Experimental): 12 week group 3 week modules: 1) Mindfulness 2) Emotion Regulation 3) Distress Tolerance
  Interventions: Behavioral: Enhancing Emotion Regulation

INTERVENTIONS:
Behavioral: Enhancing Emotion Regulation — 12 week of group therapy 3 modules: 1) mindfulness, 2) emotion regulation, 3)distress tolerance

SUMMARY:
Psychoeducation has been the only group treatment developed for bipolar disorder thus far. Deficits in emotion regulation, a core impairment among patients with bipolar disorder, are not directly addressed in this treatment. The objective of this study is to develop a group treatment for bipolar disorder that focuses on emotion regulation strategies (Enhancing Emotion Regulation; EER). This study will examine the efficacy of this treatment using an open trial design. It is hypothesized that patients who receive EER will show a reduction in mood symptoms and improvement in well-being. Reductions in emotion regulation difficulties will predict improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of bipolar I disorder.
2. Able to provide written informed consent.
3. Men or women aged 18-65.
4. Able to read and understand English.
5. Psychiatrist prescribing mood-stabilizing medication.
6. Participates in bimonthly individual psychotherapy

Exclusion Criteria:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
2. History of seizure disorder, brain injury, any history of known neurological disease (multiple sclerosis, degenerative disease such as ALS, Parkinson disease and any movement disorders, etc).
3. History or current diagnosis of the following Diagnostic and Statistical Manual of Mental Disorders, Fourth edition (DSM-IV) psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, major depressive disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 12 months.
4. Patients who currently meet criteria for a major depressive episode, a manic episode, or a mixed episode. Excluded participants may remain on a waiting list to partake in a future group dependent on mood stabilization.
5. Patients who have had electroconvulsive therapy (ECT) within the 6 months preceding enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-07; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Deckersbach, Ph.D., Principal Investigator — Bipolar Clinic and Research Program
Locations (1):
- Bipolar Clinic and Research Program, Boston, Massachusetts, United States